CLINICAL TRIAL: NCT01334463
Title: Executive Dysfunction and Self-Harm Behavior: An Examination of Veterans With Traumatic Brain Injury, Post Traumatic Stress Disorder, or Both
Brief Title: Executive Dysfunction and Self-Harm Behavior: An Examination of Veterans With TBI, PTSD, or Both
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: Colorado Traumatic Brain Injury Trust Fund (Other); University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0502
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Traumatic Brain Injury; Post Traumatic Stress Disorder; Suicide; Self-Injurious Behavior
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- mTBI+PTSD: History of active duty-related mild TBI and history of active duty-related PTSD
- mTBI Only: History of active duty-related mild TBI and no history of active duty-related PTSD
- PTSD Only: No history of active duty-related mild TBI and history of active duty-related PTSD
- No mTBI, No PTSD: No history of active duty-related mild TBI and no history of active duty-related PTSD

SUMMARY:
1. To determine whether tasks taken from the field of cognitive neuroscience can detect and distinguish impairments in executive function above and beyond standard neuropsychological measures in individuals with: a.) Mild Traumatic Brain Injury (TBI), b.) Post Traumatic Stress Disorder (PTSD), c.)Mild TBI+PTSD
2. To determine whether performance on these tasks is linked to pertinent psychiatric outcomes (e.g. history of suicidality), which is associated with compromised executive function and impulsivity.
3. To determine whether information regarding brain anatomy can provide additional information above and beyond behavior performance in distinguishing between these two groups.

DETAILED DESCRIPTION:
Individuals who served in Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) are reporting histories of traumatic brain injury (TBI) and symptoms associated with post traumatic stress disorder (PTSD). Standard neuropsychological measures are ineffective at distinguishing between TBI and PTSD. This pilot project will examine whether methods from cognitive neuroscience can determine the effects of TBI and/or PTSD on executive function. Executive function includes many aspects of goal-oriented behavior, including the ability to inhibit inappropriate behaviors and thoughts. In the proposed study, the investigators are focusing on inhibitory processing, as it is a core component of executive function. Although both TBI and PTSD compromise executive function and TBI often occurs in the context of a traumatic event, very little research has attempted to disentangle the effects that each of these conditions has on inhibitory control. In addition, the investigators are interested in how disinhibition may be linked to impulsive real-world behaviors, such as suicidal tendencies, which are observed at elevated rates in individuals with TBI as well as those with PTSD. Knowing the ways in which inhibitory functions are compromised in these individuals should aid in the development of appropriate treatments aimed at functional improvement for those with mild TBI, PTSD, or mild TBI+PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45 years old
* At least one OEF/OIF deployment
* Currently receiving or eligible to receive physical and/or mental health care through the VA Eastern Colorado Health Care System

Exclusion Criteria:

* History of other significant neurological disease (other than mild TBI for the appropriate groups) as assessed by interview and chart review
* History or diagnosis of lifetime moderate or severe TBI for the TBI groups, or any history of TBI for the non-TBI groups, as assessed by interview and chart review
* History or diagnosis of non-active duty-related mild TBI or PTSD disorder as assessed by interview and/or chart review
* Diagnosis of schizophrenia or bipolar I disorder as assessed by interview and/or chart review
* Computerized Assessment of Response Bias (CARB) performance categorized as Very Poor or Symptom Exaggerator
* Problematic drinking behavior that consistently exceeds recommended drinking limits per day, e.g., Diagnosis of Alcohol Abuse Disorder or Alcohol Dependence Disorder per the SCID; or five or more alcoholic drinks per day, four out of seven days per week for the previous two weeks
* Use of illicit substance(s) more than five times in the two weeks before enrollment
* Inability to read the informed consent document or adequately respond to questions regarding the informed consent procedure
* Contraindication to having an MRI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants in this observational study will be recruited from the following populations of OEF/OIF Veterans: 1.) those seeking mental health, rehabilitative, psychological or other services within the Veterans Health Administration (VHA) Eastern Colorado Healthcare System , 2.) those in existing clinical and research databases, and 3.) Veterans in the community not seeking care within the VHA.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2010-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Iowa Gambling Test | One time

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, Ph.D., Principal Investigator — VA Office of Research and Development
Locations (1):
- Denver VA Medical Denver, Denver, Colorado, United States